CLINICAL TRIAL: NCT05797701
Title: An Open-label, Randomized, 2-sequence, 2-period, 2-treatment, 2-part Study to Evaluate the Relative Bioavailability of SAR443820 in Tablet Formulation Versus Capsule Formulation in Fasted Condition (Part 1) and the Food-effect on SAR443820 in Tablet Formulation (Part 2) in Healthy Adult Male and Female Participants
Brief Title: A Study in Healthy Adult Male & Female Participants to Assess the Amount of the Study Medicine (SAR443820) Absorbed by the Body, When Given Orally in Fasted Condition as a Tablet Versus as a Capsule (Part 1) and When Given Orally as a Tablet in Fasted Condition Versus as a Tablet After Food (Part 2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BDR16957; U1111-1256-9220 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03-22

CONDITIONS: Amyotrophic Lateral Sclerosis (Healthy Volunteers)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): Single dose of SAR443820 tablet in fasted condition
  Interventions: Drug: SAR443820
- Treatment B (Experimental): Single dose of SAR443820 capsule in fasted condition
  Interventions: Drug: SAR443820
- Treatment C (Experimental): Single dose of SAR443820 tablet in fasted condition
  Interventions: Drug: SAR443820
- Treatment D (Experimental): Single dose of SAR443820 tablet in fed condition
  Interventions: Drug: SAR443820

INTERVENTIONS:
Drug: SAR443820 — Tablet by oral administration
  Arms: Treatment A; Treatment C; Treatment D
Drug: SAR443820 — Capsule by oral administration
  Arms: Treatment B

SUMMARY:
Part 1:

This is an open label, balanced randomized, single dose, 2-sequence, 2-period (period 1 and period 2), 2-treatment crossover (between Treatment A and Treatment B for Part 1), study part to determine the relative bioavailability of SAR443820 in tablet formulation versus capsule formulation under fasted conditions.

Two treatments are as follows:

* Treatment A: SAR443820 - tablet formulation in fasted condition
* Treatment B: SAR443820 - capsule formulation in fasted condition Each administration will be a single dose of SAR443820 separated by a wash out of at least 5 days.

Part 2:

This is an open-label, balanced randomized, single dose, 2-sequence, 2-period (period 1 and period 2), 2-treatment crossover (between Treatment C and Treatment D for Part 2) study part to perform a preliminary assessment of the effect of a high-fat meal on pharmacokinetic parameters of single dose of SAR443820 in tablet formulation.

Two treatments are as follows:

* Treatment C: SAR443820 - tablet formulation in fasted condition
* Treatment D: SAR443820 - tablet formulation in fed condition Each administration will be a single dose of SAR443820 separated by a wash out of at least 5 days.

Participants are not allowed to participate in more than one part of the study. In both Parts 1 and 2, the assessment of pharmacokinetic, safety and tolerability are performed at each treatment period at baseline (prior single dosing) up to 48-hour postdosing in healthy adult male and female participants.

DETAILED DESCRIPTION:
Screening period: up to 4 weeks (Day -28 to Day -2). In both Part 1 and Part 2: Period 1: Day -1 to Day 3 and 5 days wash out period. Period 2: Day -1 to Day 3 and until end-of-study visit at Day 6.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, body mass index between 18.0 and 30.0 kg/m^2, inclusive
* All contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Having given written informed consent prior to undertaking any study-related procedure

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of hormonal contraception or menopausal hormone replacement therapy; any non-live Covid-19 vaccine within the last 2 weeks before randomization, any live attenuated vaccine within the last 28 days before randomization and any other non-vaccine biological drugs given within 4 months before randomization
* Positive result for hepatitis B, C or human immunodeficiency virus (HIV)
* Positive result on urine drug screen
* Positive urine alcohol test
* Positive severe acute respiratory syndrom coronavirus 2 (SARS-CoV-2) test
* Any consumption of citrus fruits (grapefruit, orange, etc) or their juices within 5 days before inclusion

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum plasma concentration observed (Cmax) | In both Period 1 and Period 2: From Day 1 to Day 3
Part 2: Maximum plasma concentration observed (Cmax) | In both Period 1 and Period 2: From Day 1 to Day 3
Part 1: Area under the plasma concentration from time zero to the last concentration above the limit of quantification (AUClast) | In both Period 1 and Period 2: From Day 1 to Day 3
Part 2: Area under the plasma concentration from time zero to the last concentration above the limit of quantification (AUClast) | In both Period 1 and Period 2: From Day 1 to Day 3
Part 1: Area under the plasma concentration (AUC) | In both Period 1 and Period 2: From Day 1 to Day 3
Part 2: Area under the plasma concentration (AUC) | In both Period 1 and Period 2: From Day 1 to Day 3

SECONDARY OUTCOMES:
Part 1: Number of participants with treatment emergent adverse events (TEAEs) | In both Period 1 and Period 2: From Day 1 to Day 4
Part 2: Number of participants with treatment emergent adverse events (TEAEs) | In both Period 1 and Period 2: From Day 1 to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Prism Research-Site Number:8400001, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org